CLINICAL TRIAL: NCT00893776
Title: The Effectiveness of Bilateral Versus Unilateral Task Retraining Using the SaeboFlex Orthosis in Individuals With Subacute and Chronic Stroke.
Brief Title: Bilateral Versus Unilateral Task Retraining Using the SaeboFlex Orthosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient time for study extenuating personal circumstances of PI
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1134397
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Unilateral Group (Active Comparator): This group will wear the SaeboFlex orthosis on their affected extremity and do exercises with that extremity only. SaeboFlex exercises include moving the ball in high repetition of grasp and release while wearing the SaeboFlex orthosis to various positions individualized to each participant based on movement deficits, as well as Task Training (using the affected arm during specific functional activities to use newly acquired movement patterns)
  Interventions: Other: Task Training
- 2 Bilateral training (Experimental): Members of this group will wear the SaeboFlex orthosis on the affected extremity and do exercises with the affected extremity and the non-affected extremity at the same time. SaeboFlex exercises include moving the ball in high repetition of grasp and release while wearing the SaeboFlex orthosis to various positions individualized to each participant based on movement deficits, as well as Task Training (using the affected arm during specific functional activities to use newly acquired movement patterns)
  Interventions: Other: Task Training

INTERVENTIONS:
Other: Task Training — Task training is the movement of balls in an individually prescribed fashion using the SaeboFlex orthosis on the affected extremity.

SUMMARY:
A small, pilot study consisting of twelve participants with subacute (6-12 months post-stroke)and chronic stroke (1year+ post-stroke)living in and around Columbia area. The twelve participants will randomly be selected to participate in either unilateral (one-handed) task training (6 participants) or bilateral (two-handed) task training (6 participants) with the SaeboFlex orthosis. Each group will undergo six assessments to establish pre-testing baseline and qualification, followed by a training session, four-week combined home and clinic program, and post-testing to determine changes in affected arm use and function. The hypothesis is that two-handed training will before effective than one-handed training.

DETAILED DESCRIPTION:
The SaeboFlex device is a mechanical orthosis that promotes grasp and release and functional movement of an upper limb that has impaired movement due to a stroke. Many researchers have found that incorporating both the affected and unaffected limb together during exercises (bilateral task training) results in increased functional use of the affected limb as compared to only performing exercises with the affected limb. Therefore, we want to determine if bilateral task training is more effective than unilateral task training with the use of the SaeboFlex device in subacute and chronic stroke rehabilitation. For the unilateral training group, exercises will be completed with only the affected hand using the Saebo device. For the bilateral group, the Saebo will be on the affected hand, no device on the unaffected hand, and both arms will do the exact same movements/exercises at the same time. The participants will be videotaped and photographed moving balls without the device, with the device at the start of the study, with the device midway through the study, and at the end of the study. This will be done for the purpose of providing participant feedback regarding their progress and for report of outcomes upon completion of the project. Faces will be omitted from all photographic media at the request of the participant, and the participant may decline photographic media at any time without having to withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* >6 months post stroke
* diagnosis of first stroke
* medically stable
* ability to follow multipart verbal directions
* score of >26 on Mini-Mental Status Exam
* achieve 10 degrees elbow flexion
* 1/4 range volitional finger flexion when hand positioned in wrist and finger extension
* capable of standing for >2 minutes without an assistive ambulatory device
* maintain independence in self-care or have a caretaker to provide assistance
* no concurrent skilled therapy treatment
* not participating in any experimental rehabilitation or drug studies.

Exclusion Criteria:

* more than one stroke/multiple strokes
* receptive aphasia
* medically documented dementia
* score less than 26 on Mini Mental Status Exam
* contractures or joint deformities in the affected hand or wrist that impede the ability to use the device
* inability to transfer 12 balls crate right and 12 balls crate left, while using the Saeboflex device on the affected arm, by the end of a 5-day training session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test (WMFT) | Before and immediately after intervention

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | Before and immediately after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Giulianne Krug, MA, OTR/L, Principal Investigator — University of Missouri, Occupational Therapy and Occupational Science
Locations (1):
- University of Missouri, Lewis and Clark Hall, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This is the device we are using for the study. — http://www.saebo.com